CLINICAL TRIAL: NCT01069848
Title: Feasibility Study of the Vedera KXS for Treatment of Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Avedro T4
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Vedera KXS (Experimental)
  Interventions: Device: Vedera KXS

INTERVENTIONS:
Device: Vedera KXS — One treatment session with Vedera KXS

SUMMARY:
The objective of this investigation is to evaluate the feasibility, safety and efficacy of the Vedera KXS for the reduction or elimination of myopia and astigmatism in patients with keratoconus, who are no longer able to achieve adequate vision with their contact lenses or glasses.

ELIGIBILITY:
Inclusion Criteria:

1. 14 years of age or older
2. Presence of central or inferior steepening on the Pentacam map
3. Axial topography consistent with keratoconus
4. I-S ratio > 1.5 on the Pentacam map or topography map
5. BSCVA worse than 20/20 (<53 letters on ETDRS chart)
6. Contact Lens Wearers Only: Removal of contact lenses for the required period of time prior to the screening refraction
7. Signed written informed consent
8. Willingness and ability to comply with schedule for follow-up visits

Exclusion Criteria:

1. Eyes classified as either normal or atypical normal on the keratoconus severity grading scheme.
2. A history of previous corneal surgery or the insertion of Intacs in the eye(s) to be treated.
3. Corneal pachymetry <400 microns at diameter to be treated.
4. Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example:

   1. History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, corneal melt, corneal dystrophy, etc.)
   2. Clinically significant corneal scarring in the treatment zone that is not related to keratoconus or, in the investigator's opinion, will interfere with the treatment.
5. A history of chemical injury or delayed epithelial healing in the eye(s) to be treated.
6. Diagnosed with autoimmune disease, systemic connective tissue diseases or atopic syndrome, diabetes mellitus, or taking systemic medications likely to affect wound healing.
7. Women who are pregnant or nursing or who plan to become pregnant over the course of their participation in this investigation.

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The reduction in Kmax (by keratometry) of >1 D | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beyoglu Eye Hospital, Istanbul, Turkey (Türkiye)